CLINICAL TRIAL: NCT02553902
Title: Economic Evaluation of Treatment Modalities for Position Dependent Obstructive Sleep Apnea Patients
Brief Title: Economic Evaluation of Treatment Modalities for Position Dependent Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, L.B.L. Benoist, Drs., Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL52032.029.15
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Positional Obstructive Sleep Apnea
Keywords: Positional therapy; MAD; Oral appliance; Sleep position trainer; POSA
MeSH Terms: interventions — Occlusal Splints; Magnetic Resonance Angiography; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy (Active Comparator): Sleep Position Trainer + Mandibular Advancement device combination The SPT is a sensor that measures the sleeping position, and gives the user feedback about wrong positions with a soft vibration. A user is then able to react to the signal and turn into a non-supine position. To stimulate compliance, information is provided about nightly behaviour, implicating a learning pattern by viewing the data on a home computer.
  MRA or oral appliances (OA) works by advancing the mandible and its attached soft tissue structures forward they aim to increase upper airway size.
  Interventions: Device: Sleep position trainer; Device: Mandibular advancement device
- CPAPContinuous positive airway pressure (Active Comparator): Continuous positive airway pressure (CPAP) functions as a pneumatic splint to maintain upper airway patency. Possible side effect can be related to the interface, pressure and negative social factors.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Sleep position trainer
  Arms: Combination therapy
Device: Mandibular advancement device
  Other Names: MRA, MAD
  Arms: Combination therapy
Device: Continuous positive airway pressure
  Arms: CPAPContinuous positive airway pressure

SUMMARY:
OBJECTIVES:

To evaluate the effect and cost-utility of a combination therapy of SPT+MAD compared with continuous positive airway pressure (CPAP) in patients with moderate positional obstructive sleep apnea (POSA).

HYPOTHESIS:

The SPT+MAD combination is more cost-effective and effective, in means of reduction of the apnea-hypopnea index (AHI), quality of life and compliance, compared with CPAP.

STUDY DESIGN:

A multicenter randomized clinical trial (RCT) will be performed with a follow-up of 12 months per patient. Patients will be randomized for CPAP or the combination SPT and MRA. All outcomes will be measured at baseline, month 3, 6 and 12.

STUDY POPULATION:

Patients diagnosed with moderate POSA according to polysomnography (PSG) results.

INTERVENTION / STANDARD INTERVENTION TO BE COMPARED TO:

The SPT trains POSA patients to sleep in non-supine positions, CPAP uses positive airway pressure to open the airway; MRA is an intra-oral prosthesis, which holds the mandible in a protrusive position, all to prevent effectively apneic events.

OUTCOME MEASURES:

AHI, compliance, quality-adjusted life year (QALY), direct and indirect costs, cardiovascular parameters, incremental cost-effectiveness ratio (ICER)

SAMPLE SIZE / DATA ANALYSIS:

100 subjects in each treatment group, total of 200 patients.

COST-EFFECTIVENESS ANALYSIS / BUDGET IMPACT ANALYSIS:

The SPT is expected to improve the cost-effectiveness of overall treatment of POSA patients, and will save annually approximately 35-150 million euros.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Ability to speak, read and write Dutch
* Ability to follow up
* Diagnosis with symptomatic moderate OSA (15 < AHI < 30)
* Diagnosis of 10 to 90% supine position during the night
* AHI supine is 2 > as high as AHI non-supine
* Own a Windows PC and ability to install SPT connection software and upload research data
* Expected to maintain current lifestyle (sports, medicine, diet etc.)

Exclusion Criteria:

* Many dental problems; insufficient teeth for wearing MRA
* Medication used/ related to sleeping disorders
* Central Sleep Apnea Syndrome
* Night or shifting work
* Severe chronic heart failure
* Medical history of known causes of tiredness by day or severe sleep disruption (insomnia, PLMS, Narcolepsy)
* Seizure disorder
* Known medical history of mental retardation, memory disorders or psychiatric disorders
* Shoulder, neck and back complaints
* Reversible morphological upper airway abnormalities (e.g. enlarged tonsils)
* Inability to provide informed consent
* Simultaneous use of other treatment modalities to treat OSA
* Previous treatment for OSA with MRA, CPAP or SPT
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | change from baseline, after 3, 6 and 12 months

SECONDARY OUTCOMES:
Outcome of Quality of Life questionnaires | change from baseline, after 3, 6 and 12 months
  EQ-5D
Outcome of Quality of Life questionnaires | change from baseline, after 3, 6 and 12 months
  Epworth Sleeping Scale (ESS)
Outcome of Quality of Life questionnaires | change from baseline, after 3, 6 and 12 months
  Functional Outcome Sleep Questionnaire (FOSQ)
(Societal) costs of treatment | change from baseline, after 3, 6 and 12 months
  iMTA Productivity Cost Questionnaire (iPCQ)
(Societal) costs of treatment | change from baseline, after 3, 6 and 12 months
  iMTA Medical Consumption Questionnaire (iMCQ)
Therapy compliance | change from baseline, after 3, 6 and 12 months
  Measurement of actual wearing time (in hours) per night
Cardiovascular parameters | change from baseline, after 3, 6 and 12 months
  Systolic and diastolic blood pressure
Cardiovascular parameters | change from baseline, after 3, 6 and 12 months
  Pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: O.M. Vanderveken, Professor, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Antwerp University Hospital (UZA), Antwerp, Belgium
- OLVG West, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No